CLINICAL TRIAL: NCT04393129
Title: Prevalence of Central Sensitization Symptoms and Psychosocial Factors in Athletes After ACL Reconstruction and Return to Play
Brief Title: Central Sensitization Symptoms and Psychosocial Factors in Athletes After ACL Reconstruction
Status: Completed | Type: Observational
Sponsor: University of Thessaly (Other)
Collaborators: KAT General Hospital (Other)
Responsible Party: Principal Investigator, Eleni Kapreli, Professor, University of Thessaly
Other Study IDs: 2
Record Dates: First submitted 2020-05-08; First posted 2020-05-19 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Return to play; Psychosocial; Central sensitization; Chronic pain; Athlete; Reconstruction; Rehabilitation
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Chronic Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The main research objective of this study is whether athletes who have sustained an anterior cruciate ligament injury, experience chronic nociplastic pain and psychosocial factors, including kinesiophobia and pain catastrophizing, after having been through ACL reconstruction surgery and rehabilitation and have returned to sport.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study. For the purposes of the study a sample group was selected from a clinic specialised in ACL reconstruction and rehabilitation based in Athens, Greece. Patients of the specific clinic had received the same surgical technique and rehabilitation protocol. Ability to return to sport was examined 9 months after surgery and approval was given according to the rehabilitation progress. A list of eligible study subjects was formed and, after inclusion and exclusion criteria were screened for, they were invited to participate in the study. Study participants, after having declared consent and passed the criteria were asked to answer the study questionnaires. Communication with participants was done through telephone and email, and all questionnaires were completed online.

ELIGIBILITY:
Inclusion Criteria:

1. knowledge of Greek language,
2. surgically reconstructed ACL tear on one limb only,
3. successful completion of rehabilitation program,
4. medical permission to return to sport,
5. returned to previous sport for at least 6 months period
6. athlete of a lower limb loading sport.

Exclusion Criteria:

1. adolescent age (<18 years of age),
2. diagnosis of cancer of any stage,
3. diagnosis of psychiatric, neurological or autoimmune disease or syndrome,
4. past musculoskeletal injuries, including fractures, joints dislocation, ligament and tendon tears and
5. chronic musculoskeletal injuries (tendinopathies, shin splints, shoulder impingement etc.). Chronic pain is defined as pain persisting for at least 3 months, of intensity at least 3 on the VAS scale for most days per week (Kuppens et al. 2018).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Athletes that have suffered an ACL rupture and have undergone surgical reconstruction and rehabilitation, and have been cleared to return to sport.
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-03-05 (Actual)

PRIMARY OUTCOMES:
Symptoms of Central Sensitization | At least 9 months post-operative
  The Central Sensitization Inventory (CSI) was used to assess symptoms of central sensitization. CSI was developed as a tool to evaluate somatic and emotional complaints associated with central sensitization syndrome. The CSI consists of 25 questions and can be divided in four sections that focus on physical symptoms, emotional distress, headache and jaw symptoms and urological symptoms (Mayer et al. 2012). Each question is answered on a 0-4 scale by choosing the intensity that best describes their symptoms or emotions. The individual answers are added to form a total score that can range from 0 to 100.
Pain intensity | At least 9 months post-operative
  The Numerical Rating Scale (NRS) was used to assess pain intensity. NRS has been widely used to measure and assess pain levels in adults, including chronic pain patients (Hawker et al. 2011). The scale consists of a segmented numeric version of the Visual Analog Scale (VAS) in which subjects choose a number (0-10) that best describes their pain intensity.
Pain Catastrophizing | At least 9 months post-operative
  Pain catastrophizing was assessed by the Pain Catastrophizing Scale (PCS). PCS was created in an effort to measure inability to cope with pain due to catastrophizing. The scale was developed on the construct that catastrophizing involves three subsequent dimensions, rumination, magnification and helplessness (Craner et al. 2016). It is a self-report questionnaire which includes 13 items about the above three dimensions of pain catastrophizing. Every item is answered on a Likert scale ranging from 0 to 4. A final total score will range between 0 and 52 points with minimal detectable change being 9 points.
Kinesiophobia | At least 9 months post-operative
  Kinesiophobia was assessed using the Tampa Scale for Kinesiophobia (TSK). TSK is a questionnaire which consists of 17 questions and is used to assess fear of movement and re injury. The questions are answered by choosing the statement that most accurately represents the subjects state, these answers vary from "strongly agree" to "strongly disagree". The final score of the questionnaire will range from 17-68 and is made up by scoring each answer in a Likert scale (Lundberg et al. 2011).
Sense of unfairness | At least 9 months post-operative
  Sense of unfairness was examined by using the Inequality Experience Questionnaire (IEQ) which is a 12-item scale that asks participants to indicate the frequency with which they experience different thoughts concerning the sense of unfairness corelated to their injury on a five-point scale ranging from 0 (never) to 4 (all the time). The IEQ yields two factors that have been labeled severity/irreparability of loss and blame/unfairness. The IEQ has been shown to be internally reliable (Sullivan et al. 2008).
  The IEQ total score is measured by summing responses to all 12 items.
Illness Perception | At least 9 months post-operative
  Brief Illness Perception Questionnaire (B-IPQ) was used to assess illness perception. The B-IPQ is a very commonly used tool to assess the subject's perception of their illness. In total it consists of 9 items which are scored on a 0-10 scale apart from the final item which is an open-ended question.

SECONDARY OUTCOMES:
Willingness and ability to return to play | At least 9 months post-operative
  Anterior Cruciate Ligament - Return to Sport after Injury (ACL-RSI) questionnaire was used to assess willingness and ability to return to play. The ACl-RSI scale focuses on three main psychosocial areas, emotions, confidence and risk appraisal, that can affect willingness and ability to return to sport safely. The scale has high internal consistency, Cronbach's alpha 0.96 and inter-item correlations were high with a mean of 0.69 (min 0.49, max 0.83) (Webster et al. 2008). The ACL-RSI consists of a unidimensional 12-question scale that measures the three psychosocial domains mentioned above, 5 questions focus on emotions, 5 on confidence in performance and 2 on risk appraisal. The questions are answered on a scale from 0 to 100 in 10-point increments and the total score is represented by the mean total of the answers' given (Webster et al. 2008).
Activity level | At least 9 months post-operative
  Tegner Activity Scale (TAS) was used to assess the activity level. Activity level and level of sports participation of athletes recovering from ACL is most often measured by self-report and the Tegner Activity Scale (TAS) or by a combination of the above (Neeb et al. 1997). The TAS is a grades activity based on work and sport activities. The TAS consists of a numerical scale (0-10) followed by a sentence describing each level of activity. The subjects is asked to choose the number that best describes their activity level. A higher score indicates a higher activity level. Test retest validity has been found to be acceptable (ICC> 0.70) and internal validity was measured to be a=0.72 (Cronbach). Specifically, the TAS has been tested in the ACL population and seems to demonstrate acceptable psychometric parameters (Briggs et al. 2009).
Knee functional level | At least 9 months post-operative
  Knee injury and Osteoarthritis Outcome Score (KOOS) was used to assess knee functional level. It is a knee specific measuring instrument which was originally developed in order to evaluate both the short-term and long-term consequences of a knee injury. The KOOS questionnaire consists of five subgroups referring to pain, symptoms, activities of daily living, sports and recreation functionality and quality of life. In total there are 42 questions and It has been validated on the anterior cruciate ligament reconstruction population and is considered most appropriate for this study since it assesses sport and recreation functionality (Roos and Lohmander 2003).

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Kapreli, Phd, Study Chair — Physiotherapy Department, University of Thessaly
Locations (1):
- Clinical Exercise Physiology and Rehabilitation Laboratory, Lamia, Central Greece, Greece

REFERENCES:
- [Background] Craner JR, Gilliam WP, Sperry JA. Rumination, Magnification, and Helplessness: How do Different Aspects of Pain Catastrophizing Relate to Pain Severity and Functioning? Clin J Pain. 2016 Dec;32(12):1028-1035. doi: 10.1097/AJP.0000000000000355. PMID 26783987
- [Background] Kuppens K, Hans G, Roussel N, Struyf F, Fransen E, Cras P, Van Wilgen CP, Nijs J. Sensory processing and central pain modulation in patients with chronic shoulder pain: A case-control study. Scand J Med Sci Sports. 2018 Mar;28(3):1183-1192. doi: 10.1111/sms.12982. Epub 2017 Oct 4. PMID 28980347
- [Background] Lundberg M, Grimby-Ekman A, Verbunt J, Simmonds MJ. Pain-related fear: a critical review of the related measures. Pain Res Treat. 2011;2011:494196. doi: 10.1155/2011/494196. Epub 2011 Nov 15. PMID 22191022
- [Background] Mayer TG, Neblett R, Cohen H, Howard KJ, Choi YH, Williams MJ, Perez Y, Gatchel RJ. The development and psychometric validation of the central sensitization inventory. Pain Pract. 2012 Apr;12(4):276-85. doi: 10.1111/j.1533-2500.2011.00493.x. Epub 2011 Sep 27. PMID 21951710
- [Background] Roos EM, Lohmander LS. The Knee injury and Osteoarthritis Outcome Score (KOOS): from joint injury to osteoarthritis. Health Qual Life Outcomes. 2003 Nov 3;1:64. doi: 10.1186/1477-7525-1-64. PMID 14613558
- [Background] Sullivan MJ, Adams H, Horan S, Maher D, Boland D, Gross R. The role of perceived injustice in the experience of chronic pain and disability: scale development and validation. J Occup Rehabil. 2008 Sep;18(3):249-61. doi: 10.1007/s10926-008-9140-5. Epub 2008 Jun 7. PMID 18536983
- [Background] Webster KE, Feller JA, Lambros C. Development and preliminary validation of a scale to measure the psychological impact of returning to sport following anterior cruciate ligament reconstruction surgery. Phys Ther Sport. 2008 Feb;9(1):9-15. doi: 10.1016/j.ptsp.2007.09.003. Epub 2007 Nov 5. PMID 19083699